CLINICAL TRIAL: NCT06947811
Title: A Multicenter, Open-Label, Single-Arm, Phase Ib/II Clinical Study of Almonertinib Combined With Palbociclib in the Treatment of Patients With KRAS Mutations-Positive Advanced Solid Tumors
Brief Title: A Study of Almonertinib Combined With Palbociclib in Patients With Advanced Solid Tumors Harboring KRAS Mutations
Acronym: APEAK
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hongyun Zhao, Associate Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-058
Record Dates: First submitted 2025-04-14; First posted 2025-04-27 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: EGFR Tyrosine Kinase Inhibitors Plus Cyclin-dependent Kinase 4/6 Inhibitor
Keywords: EGFR Tyrosine Kinase Inhibitors; Cyclin-dependent kinase 4/6 inhibitor; solid tumor
MeSH Terms: interventions — aumolertinib; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Almonertinib + Palbociclib (Experimental): Part 1: Phase I open-label dose-escalation study. The dose of Ameitinib (110mg) remains unchanged, while the administration frequency of palbociclib will be adjusted based on patient tolerance. Dosing regimen: Palbociclib capsules 125mg, orally once daily (qd) for 21 consecutive days followed by a 7-day break + Ameitinib 110mg, orally once daily (qd); administered on an empty stomach, with each treatment cycle lasting 4 weeks.
  Part 2: Single-arm Phase II clinical study, based on the dosing regimen of palbociclib capsules determined during the safety run-in phase. Dosing regimen: Palbociclib capsules 125mg, orally once daily (qd), administered on an empty stomach for 21 consecutive days followed by a 7-day break (tentative) + Ameitinib 110mg, orally once daily (qd), administered on an empty stomach for 28 consecutive days; each treatment cycle lasts 4 weeks.
  Interventions: Drug: Almonertinib; Drug: Palbociclib

INTERVENTIONS:
Drug: Almonertinib — Patients will be treated with Almonertinib, 110 mg p.o., daily
Drug: Palbociclib — Patients will be treated with Palbociclib, 125 mg(dose determined from Part one of study) p.o., daily

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of almonertinib combined with palbociclib in patients with advanced solid tumors harboring KRAS gene mutations, and to conduct a preliminary observation of its efficacy

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the safety and tolerability of almonertinib combined with palbociclib in patients with advanced solid tumors harboring KRAS gene mutations, and to conduct a preliminary observation of its efficacy

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 70 years of age (containing threshold levels), no gender restrictions.
2. Eastern Cooperative Oncology Group (ECOG) performance scale 0 - 1.
3. Life expectancy of no less than 12 weeks. Histologically or cytologically confirmed advanced solid tumors (including but not limited to lung cancer, pancreatic cancer, colorectal cancer, etc.),who meet at least one of the following criteria：

   * tissue and/or ctDNA samples with KRAS mutation (including but not limited to G12C，G12D，G13D，G12V，G12S, etc.) .
   * failure of prior standard therapy or no standard treatment is available.
4. Any toxicities related to prior anticancer therapy must have recovered to ≤ Grade 1 (excluding alopecia).
5. Have not received chemotherapy or other targeted therapies previously.

   -note: Therapies administered during the neoadjuvant treatment phase are not counted as prior treatment regimens; patients who experience disease recurrence within 6 months after completion of adjuvant therapy will have the adjuvant therapy considered as first-line therapy and are not eligible for this study; for recurrence occurring >6 months after completion of adjuvant therapy, the adjuvant therapy will not be counted as a prior treatment regimen.
6. Patients who have received prior radiotherapy are eligible for enrollment, provided that: the irradiated area involves <25% of the bone marrow (Cristy and Eckerman 1987), and no whole pelvic or thoracic irradiation has been administered; prior radiotherapy must have been completed at least 4 weeks before study enrollment, any acute toxicities related to previous radiotherapy must have resolved; previously irradiated lesions cannot be considered measurable target lesions unless documented progression is observed after the last radiotherapy session.
7. Adequate organ function prior to the first dose of the study drug, with cardiac, hematological, hepatic, and renal functions meeting protocol-specified requirements as defined by the following criteria:

   * Hematological laboratory tests must meet the following criteria:

     1. ANC≥1.5×109/L；
     2. PLT≥100×109/L；
     3. Hb≥100g/L.
   * The biochemical examination must meet the following criteria:

     1. TBIL<1.5×ULN；
     2. ALT、AST and ALP<2.5×ULN；
     3. BUN and Cr≤1×ULN or endogenous creatinine clearance rate≥50ml/min（Cockcroft-Gault formula）.
8. Female subjects of childbearing potential must have either practiced reliable contraceptive methods or undergone a pregnancy test (serum or urine) within 7 days prior to enrollment with negative results, and must be willing to use appropriate contraceptive methods during the trial period and for 8 weeks after the last administration of the investigational drug. Male subjects must agree to use appropriate contraceptive methods during the trial period and for 8 weeks after the last administration of the investigational drug, or have been surgically sterilized.
9. Subjects must voluntarily participate in the study, sign an informed consent form, demonstrate good compliance, and actively cooperate with follow-up procedures.
10. Subjects are requested to provide, whenever possible, previous tumor tissue paraffin blocks (or 5-15 pathological biopsy sections [unstained slides]) and peripheral blood specimens (10ml), and to cooperate with investigators during treatment for tumor biopsy sampling when feasible, to support exploratory research on tumor biomarker detection.

Exclusion Criteria:

Patients presenting with any of the following criteria will be excluded from the study:

1. Exclusion applies to patients who had symptomatic CNS metastases, leptomeningeal metastases, or spinal cord compression caused by metastatic lesions prior to signing the informed consent form.
2. Patients with prior or current use of CDK4/6-targeted anticancer agents.
3. Molecular targeted therapy or radiotherapy within 2 weeks prior to screening; Chemotherapy or immunotherapy within 3 weeks prior to screening; Nitrosoureas or mitomycin administration within 6 weeks prior to screening; Prior radical radiotherapy involving ≥25% of bone marrow, inclusion eligibility subject to investigator evaluation.
4. Major surgery performed within 6 weeks prior to screening, or planned major surgery within 12 weeks after initiation of the investigational drug.
5. Patients who have participated in other clinical studies with active treatment exposure within 28 days before the first investigational drug dose are ineligible.
6. Third-space fluid accumulations refractory to drainage or therapeutic interventions exist (such as massive pleural effusions, ascites, and pericardial effusions).
7. Active inflammatory bowel disease, chronic diarrhea, intestinal obstruction, dysphagia, or the presence of multiple factors that impair drug administration and absorption.
8. Uncontrolled electrolyte disturbances (e.g., hypocalcemia, hypokalemia, hypomagnesemia).
9. Individuals with allergic predisposition or a history of severe allergic reactions.
10. Active hepatitis B virus (HBV) infection; active hepatitis C virus (HCV) infection; history of immunodeficiency.
11. Documented long QT syndrome (congenital/acquired) or familial LQTS with genetic confirmation; significant ventricular arrhythmias (e.g., sustained VT/VF), ongoing antiarrhythmic therapy, or ICD implantation; grade 3+ (CTCAE v5.0) cardio/cerebrovascular events within 6 months pre-dosing; NYHA functional class III-IV.
12. Suffers from severe lung disease (interstitial lung disease, severe chronic obstructive pulmonary disease [COPD], severe pulmonary insufficiency, and a history of symptomatic bronchospasm).
13. Pregnant or lactating women; women of childbearing potential with a positive baseline pregnancy test; and women of childbearing age or male patients with partners of childbearing age who are unwilling to use effective contraception throughout the trial period.
14. Presence of concomitant diseases deemed by the investigator to pose significant risks to patient safety or compromise study completion.
15. Documented history of neurological or psychiatric disorders, including epilepsy or dementia.
16. Other conditions deemed by the investigator to preclude safe and appropriate study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2025-06-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Safety and Tolerability Assessment : Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0 [Time Frame: Randomization to Measured Progressive Disease (Estimated as 50 Months)]
Objective Response Rate (ORR) | Objective Response Rate (ORR) [Time Frame: Randomization to Disease Progression (Estimated as 42 Months)]

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Progression Free Survival (PFS) [Time Frame: Randomization to Measured Progressive Disease or Death from Any Cause (Estimated as 42 Months)]

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No